CLINICAL TRIAL: NCT04972864
Title: Effects of Respiratory Muscle Training in Patients With Post COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fulden Sarı, Msc, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 203
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: COVID-19; inspiratory muscle training; respiratory muscle training; exercise
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training group (Active Comparator): Individuals in the treatment group were given respiratory exercises (diaphragmatic breathing, thoracic expansion, exercises to increase chest compliance with respiratory control with exercise band and leg strengthening exercises) and inspiratory muscle training with the Threshold IMT (T-IMT) device. Inspiratory muscle training was applied for 30 minutes, 3 times a day, 7 days a week for 6 weeks.
  Interventions: Other: Exercise training group
- Control training group (Placebo Comparator): Breathing exercises (diaphragmatic breathing, thoracic expansion, exercises to increase chest compliance with respiratory control with exercise band and leg strengthening exercises) were taught in the control group and only the exercise link containing these exercises was sent.
  Interventions: Other: Control training group

INTERVENTIONS:
Other: Exercise training group — A regular advanced exercise program was given and followed.
  Arms: Exercise training group
Other: Control training group — Basic exercises was given at the beginning and did the same exercises
  Arms: Control training group

SUMMARY:
The coronavirus disease 2019 (COVID-19) outbreak first appeared in Wuhan, China's Hubei Province in December 2019 and has quickly turned into a worldwide pandemic. As of 28 July 2020, 16,465,707 cases of COVID-19 have been reported. COVID-19 is a highly contagious respiratory disease that causes respiratory, physical and psychological dysfunction in patients.

Severe respiratory symptoms have been observed in COVID-19 patients. Fever (88.7%), cough (57.6%) and shortness of breath (45.6%) were observed in an average of 81% of the patients. However, patients with comorbidities such as hypertension and diabetes, usually over 65 years of age, may have very serious pulmonary sequelae of the infection. Due to lung fibrosis as a result of pneumonia in COVID-19, some patients experience severe respiratory failure requiring pulmonary rehabilitation. In the study of Complaints such as peripheral and respiratory muscle weakness, shortness of breath on exertion, and decreased exercise capacity may be seen in patients who have had COVID-19. In addition, while anxiety and depression increase, quality of life may decrease. In a study conducted with geriatric patients who had COVID-19 and were discharged; Peripheral and respiratory muscle strengthening exercises were given to the patient after discharge, and as a result of the study, it was found that the patient's walking distance and cough strength increased, while the complaints of shortness of breath, anxiety and depression decreased significantly. As a result of this; We can say that while shortness of breath, anxiety-depression and complications are reduced with the pulmonary rehabilitation program in patients with pulmonary involvement who have had COVID-19, participation in daily life activities and quality of life increase.

Telerehabilitation is an emerging method that aims to provide rehabilitation to patients and clinicians by reducing barriers such as distance, time and cost by using information and communication technologies. Telerehabilitation enables patients who cannot access rehabilitation due to geographic, economic or physical disabilities to benefit from rehabilitation services. At the same time, the importance of social distance is emphasized for the continuation of the pandemic process and protection from the highly contagious COVID-19 infection.

DETAILED DESCRIPTION:
Outpatients with pulmonary involvement who have had COVID-19 was included in the study. Patients who had COVID-19 and pulmonary problems was divided into two groups as randomized controlled. Individuals in the first group was given respiratory exercises (diaphragmatic breathing, thoracic expansion, exercises to increase chest compliance with respiratory control with exercise band and leg strengthening exercises) and inspiratory muscle training with the Threshold IMT (T-IMT) device. The T-IMT (Threshold IMT, Respironics, USA) is a device that provides the same pressure with each breath for the strength and endurance of the inspiratory muscles, regardless of whether the patient is breathing rapidly or slowly. This device provides a constant pressure during inspiration with its flow-independent one-way valve. At the same time, the tool has an adjustable pressure mechanism. The instrument consists of the pressure section, the mouthpiece and the nose clip. When the patient breathes deeply, a constant pressure is applied to inspiration by the valve and the respiratory muscles are strengthened. In the study, individuals was divided into two groups by randomization method. In the first group, inspiratory muscle training was applied for 30 minutes, 3 times a day, 7 days a week for 6 weeks. In practice, individuals was asked to sit in a relaxed upper chest and shoulders position. After the nose clip was in place, the patient was taught to inhale and exhale by closing their lips tightly around the mouthpiece of the instrument. After 8-10 breathing cycles, the patient was asked to continue this cycle for 10 minutes at a time, by checking the breathing for 3-4 breaths. The presence of symptoms such as dizziness, fatigue and shortness of breath was also questioned during the training. In the second group; only breathing exercises (diaphragmatic breathing, thoracic expansion, exercises to increase chest compliance with respiratory control with exercise band, and leg strengthening exercises) was given and a youtube video was sent to the patients so that they could follow the exercises and they was interviewed regularly every week. In the second group; breathing exercises (diaphragmatic breathing, thoracic expansion, exercises to increase chest compliance with respiratory control with exercise band and leg strengthening exercises) was taught and only the exercise link with these exercises was sent.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65
* Those with a history of COVID-19 and symptomatic pulmonary distress
* Having an acquaintance who has or knows minimum smartphone or computer usage knowledge
* Being literate

Exclusion Criteria:

* Patients who cannot cooperate with the assessment
* Those who have orthopedic problems or neurological diseases that will affect the evaluation of functional capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-07-18 (Actual)

PRIMARY OUTCOMES:
Functional exercise capacity | First day
  Functional exercise capacity was evaluated with the 6-minute walk test according to the European Respiratory Society and American Thoracic Society (ATS/ERS) criteria. Patients were asked to walk as fast as possible at their own walking pace for 6 minutes on a 30-meter straight corridor. Oxygen saturation and heart rate (Beurer pulse oximeter, Ulm, Germany), respiratory frequency, Respiratory frequency, dyspnea, fatigue and leg fatigue perception (modified Borg scale)were recorded before and after the test and during 1 minute recovery.
30 second sit and stand test | First day
  It is a test that evaluates the 30 seconds sit-to-stand activity (30 STS), lower extremity strength and dynamic balance of the patient. The number of times the patient sits and stands in 30 seconds gives the score of the test.
International Physical Activity Questionnaire-short form | First day
  Physical activity level was evaluated with Turkish valid and reliable International Physical Activity (IPAQ) questionnaire. The questionnaire consisting of 7 questions gives information about the time spent in walking, moderate-to-vigorous and vigorous activities. The time spent sitting is considered as a separate question. A score is obtained in total score metabolic equivalent (MET)-minutes. According to the result, physical activity level is classified as 'inactive', 'minimally active' and 'very active' .
Numerical Evaluation Scale-Pain | First day
  The Numeric Rating Scale (NRS) was used to determine the pain level of the patients at rest, activity and at night. Patients are asked to mark the numbers between 0 and 10 at the time of assessment, in terms of rest, activity and night pain.
Nottingham Health Profile | First day
  The assessment of quality of life was assessed with the Nottingham Health Profile (NHP). The questionnaire consists of 38 items and 6 subgroups. There is a possible score limit for each subgroups, ranging from 0-100. 0 indicates no restrictions, 100 indicates presence of all listed restrictions.
Hospital Anxiety and Depression Scale | First day
  A valid and reliable Turkish Hospital Anxiety and Depression Scale (HADS) was used to determine the anxiety and depression levels of the patients. In the questionnaire consisting of a total of 14 questions, odd-numbered questions assess anxiety and even-numbered questions assess depression. It has two subgroups, anxiety (HADS-A) and depression (HADS-D). The lowest score that patients can get from both subgroups is 0, and the highest score is 21.
Modified Medical Research Council Dyspnea Scale | First day
  Assessment of dyspnea was assessed with the Modified Medical Research Council (MMRC) dyspnea scale. The MMRC is a category scale consisting of 5 statements about dyspnea, scored between 0-4.
Fatigue Severity Scale | First day
  It was evaluated with the Fatigue Severity Scale (FSS). It is a scale used by the individual to determine the perception of fatigue. The scale consists of nine items, each item is scored between 1-7. An increase in the total score obtained from the scale indicates that the severity of fatigue of the individual increases

CONTACTS AND LOCATIONS:
Overall Officials: Deran OSKAY, Prof, Study Director — Gazi University
Locations (1):
- Gazi University, Çankaya, Ankara, Turkey (Türkiye)